CLINICAL TRIAL: NCT01921998
Title: Development of a Biomarker Directed Strategy to Ameliorate Common Toxicities From Conventional Chemotherapy
Acronym: BioACT
Status: Suspended | Type: Observational
Why Stopped: Trial has been suspended due to lack of resource and staff
Sponsor: The Christie NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Rebecca Robinson, Clinical Trial Project Manager, The Christie NHS Foundation Trust
Other Study IDs: 11_DOG05_99
Record Dates: First submitted 2013-08-09; First posted 2013-08-14 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Lymphoma; Sarcoma
MeSH Terms: conditions — Lymphoma; Sarcoma | interventions — Biomarkers; Health Care Economics and Organizations

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected to analyse for biomarkers CK18 and FLT 3 Ligand.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Biomarker and health economics: Biomarkers will be taken throughout cycle 1. Health economics will be recorded using a patient side effect diary, a details of admission form, and a patient survey of healthcare use.
  Interventions: Procedure: Biomarker and health economics

INTERVENTIONS:
Procedure: Biomarker and health economics — Biomarkers CK18 and FLT3 Ligand will be collected

SUMMARY:
Side effects from chemotherapy can be severe in some patients leading to admission to hospital, a worse quality of life and delays in subsequent doses of chemotherapy. A blood test that could predict patients who will go on to develop severe side effects could be useful and might allow early intervention with medicines to reduce the severity of the symptoms and prevent admission to hospital.

This study will collect blood samples from patients with lymphoma or sarcoma who are receiving chemotherapy (with an expected admission rate for neutropenic sepsis, one of the side effects that most commonly results in hospital admission, of less than 20%). It will assess whether changes in blood proteins ("biomarkers") taken 2 days after the 1st chemotherapy can predict subsequent severe side effects throughout the 4 months of chemotherapy. In addition the investigators will collect data on quality of life and contact with medical professionals to assess the costs of chemotherapy toxicity to both the patient and health service. This will allow us in the future to model the cost effectiveness of using biomarkers in this manner to try and reduce chemotherapy toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lymphoma or sarcoma identified to receive out-patient chemotherapy with an anticipated febrile neutropenia rate of less than 20%. This would include 21 day R-CHOP in patients under 70 and single agent doxorubicin [Aapro et al, 2011a].
* Age 18 or older
* Performance Status 0-2
* Before patient registration, written informed consent must be given according to ICH/GCP, and national regulations.

Exclusion Criteria:

* Past history of HIV, Hepatitis B or C positive, due to the difficulties in handling high-risk specimens within CEP.
* Major surgery, radiotherapy, chemotherapy or mechanism based agents within the last 4 weeks.
* Radio-immunotherapy within the last 8 weeks.
* Bilirubin greater than 1.5 X the upper limit of normal and ALT greater than 2.5 x the upper limit of normal (as disturbed liver function tests are associated with elevated CK18) [Gonzalez-Quintela et al, 2009, Lavallard et al, 2011]
* Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Lymphoma or sarcoma identified to receive out-patient chemotherapy with an anticipated febrile neutropenia rate of less than 20%.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
sensitivity and specificity of changes in CK18 and FLT 3 ligand at day 3 of chemotherapy to predict subsequent severe toxicity | day 3
  to confirm in a prospective cohort whether changes in CK18 and FLT3 ligand at day 3 of chemotherapy can identify patients at risk of subsequent severe chemotherapy toxicity

SECONDARY OUTCOMES:
number of hospital admissions for febrile neutropenia | end of chemotherapy at approximately 6 months
Total number of overnight stays or stays in A&E of over 4 hours spent in hospital | End of study chemotherapy at approximately 6 months
Dose intensity of chemotherapy achieved compared to planned cumulative dose on initiation of therapy | End of chemotherapy at approximately 6 months
Number of total days delay in receiving chemotherapy treatment compared to planned delivery | end of chemotherapy at approximately 6 months
Change in QOL at the start of cycles 2, 4 and 6 of chemotherapy and at the end of study as measured by functional assessment of cancer therapy general (FACT-G) and euroqol EQ-5D questionnaires | cycle 2 (week6), 4 (week 12), 6 (week 18) and end of study (approximately 6 months)
Total number of contacts (both face to face and telephone) with medical and nursing staff including visits to GP, Accident and Emergency, hospital clinics and telephone consultations with Hotline staff of hospital doctors | end of study chemotherapy at approximately 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Alastair Greystoke, Study Chair — The Christie NHS Foundation Trust
Locations (1):
- The Christie NHS Foundation Trust, Manchester, United Kingdom